CLINICAL TRIAL: NCT07345949
Title: Panniculitis in Dermatomyositis
Acronym: PANNICUL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9944
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Panniculitis; Dermatomyositis
Keywords: Panniculitis; Dermatomyositis; Adipose tissue
MeSH Terms: conditions — Panniculitis; Dermatomyositis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adipose tissue involvement is rare in dermatomyositis. The occurrence of partial or diffuse lipodystrophy is a rare but well-characterized manifestation, particularly in juvenile forms of dermatomyositis. Panniculitis, on the other hand, is exceptional and rarely described in the literature, mostly in the form of clinical cases.

Panniculitis in dermatomyositis is exceptional. There are no validated diagnostic criteria or treatment recommendations. Treatment is based, by analogy, on the therapeutic strategy for lupus panniculitis and involves synthetic antimalarials combined with steroids and/or immunosuppressants.

The aim of this study is to describe panniculitis in dermatomyositis in order to determine whether there are clinical or histological characteristics that distinguish it from other causes of panniculitis, particularly panniculitis associated with lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 1 year and older
* With a confirmed diagnosis of dermatomyositis
* With a confirmed diagnosis of panniculitis

Exclusion Criteria:

* Panniculitis for which another cause has been established, particularly infectious and metabolic panniculitis

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subject with a confirmed diagnosis of dermatomyositis and panniculitis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04-20 (Estimated)

PRIMARY OUTCOMES:
Determine the clinical and histological characteristics of panniculitis in dermatomyositis | Up to 30 months
  The investigators aim to describe:
  how inflammation of the subcutaneous fat manifests
  * in individuals with dermatomyositis
  * both:
    * clinically and visually in the patient
    * under the microscope (histology)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de dermatologie - CHU de Strasbourg - France, Strasbourg, France